CLINICAL TRIAL: NCT06036459
Title: Effect of Uterine Peristalsis at the Time of Embryo Transfer on the Outcomes of IVF Cycles: a Prospective Cohort Study
Brief Title: Uterine Peristalsis in IVF
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Abdallah, Principle investigator, Assiut University
Other Study IDs: Uterine Peristalsis in IVF
Record Dates: First submitted 2023-08-13; First posted 2023-09-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: uterine peristalsis — Transabdominal us followed by Transvaginal ultrasonography scans (Sono Ace R5 ) of uterine peristalsis will performed on the day of embryo transfer while the patient lying relaxed in lithotomy position. The probe will be introduced into the vagina as gently as possible to avoid stimulating the cervix. After scanning the mid-sagittal plane of the uterus, the probe will be fixed as steady as possible while a 3 min video of uterine peristalsis will be recorded simultaneously. The records will be analyzed at 4X regular speed using a Video player application by two independent experienced observers. The uterine peristaltic wave frequency will be the mean of the results from each observer.

SUMMARY:
An observational prospective cohort study to evaluate the effect of uterine peristalsis at the time of embryo transfer on IVF clinical outcomes performed in Women's Health hospital, Assiut University, Egypt.

Women performing fresh or frozen embryo transfer who do not have any uterine abnormalities will be included in the study

ELIGIBILITY:
Inclusion Criteria:

* • Women undergoing embryo transfer during IVF cycles.

  * Age: between 20 and 40 years.
  * Have at least 1 good quality embryo at the time of transfer
  * Fresh or frozen-thawed cycles.
  * Any stimulation protocol in fresh cycles, or any endometrial preparation protocol for frozen-thawed cycles

Exclusion Criteria:

* • Women refusing to participate in clinical research.

  * Any uncorrected uterine abnormality, such as septum, myoma, adenomyosis, or polyp
  * Hydrosalpinx without prior disconnection or excision

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing IVF
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | 2 weeks after a positive pregnancy test
  The presence of intrauterine gestational sac and fetal pole with positive cardiac pulsation by transvaginal ultrasound

SECONDARY OUTCOMES:
Biochemical pregnancy | 2 weeks after embryo transfer
  a positive serum human chorionic gonadotropin
Miscarriage | From 6 weeks of gestation until 28 weeks of gestation
  Pregnancy loss either loss of cardiac pulsation by ultrasound, or spontaneous loss of pregnancy vaginally
Ectopic pregnancy | the site of the gestational sac will be assessed 2 weeks after embryo transfer
  Pregnancy outside the uterine cavity
Ongoing pregnancy | After 12 weeks of gestation until delivery
  The presence of a viable pregnancy after 12 weeks of gestation
Live birth | From 28 weeks of gestation until delivery
  Delivery of a living foetus after the age of viability

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdelaziz, M.Sc, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided